CLINICAL TRIAL: NCT06661512
Title: Acquired Brain Injury and Neurorehabilitation: the Influence of Psychological Characteristics
Acronym: DANEA
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Guttmann (Other)
Responsible Party: Sponsor
Other Study IDs: 2024431_2
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Brain Injury; Stroke Patients; TBI-Traumatic Brain Injury
Keywords: brain injury; neurorehabilitation; psychological characteristics
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic | interventions — Neurological Rehabilitation; Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Acquired Brain Injury: Any patient who begins neurorehabilitation treatment at the Institut Guttmann Neurorehabilitation Hospital (Badalona) during the recruitment period will be considered a candidate for the study. The inclusion and exclusion criteria will then be checked, and those who meet the criteria will be offered participation in the study.
  Interventions: Other: Neurorehabilitation program

INTERVENTIONS:
Other: Neurorehabilitation program — Participants will participate in a neurorehabilitation program, consisting in a structured, interdisciplinary approach designed to help individuals improve their functional abilities following acquired brain injury. The goal is to optimize the individual's physical, cognitive, emotional, and social functioning to enhance their quality of life
  The neurorehabilitation program includes, physical rehabilitation, occupational therapy, speech therapy and neuropsychological rehabilitation (cognitive, emotional and behavioral).
  Other Names: Neurorehabilitation; Rehabilitation; multidisciplinar rehabilitation

SUMMARY:
Acquired brain damage generates motor, cognitive, behavioral and emotional deficits. Neurorehabilitation aims to reduce these deficits and develop compensatory strategies that increase the person's functionality. However, the success of neurorehabilitation process varies and is influenced by the type of injury, the characteristics of the patient or the treatment received. Despite all the studies about patient characteristics, psychological aspects currently continue to be a field to be explored.

The main objective of the study is to study the psychological characteristics of people with brain damage. Secondary objectives include analyzing its link with other indicators, exploring possible differences depending on the etiology of brain damage, assessing its evolution during neurorehabilitation and exploring its prognostic value.

To carry out this prospective longitudinal observational study, adult patients with acquired brain damage to less than 6 months of evolution who present an objective cognitive alteration will be selected. Patients with a neurological or psychiatric history will be excluded.

Patients included in the study will be administered computerized questionnaires at the beginning of the neurorehabilitation program. The same questionnaires will be administered again 2 months later. In those hospitalized patients who subsequently continue outpatient treatment, a third administration will be performed (2 months after the second administration).

DETAILED DESCRIPTION:
The neurorehabilitative process can be influenced by different factors. Among the most studied are those related to the characteristics of the patient (age, level of education...), the injury (nature, location, magnitude...) or the treatment received (early, intensive...). In contrast, the possible influence of the patient's psychological characteristics on the neurorehabilitation process has been little studied.

Published research on the role of psychological characteristics in the neurorehabilitation process has focused on populations with mild brain damage, using cross-sectional methodologies. The researchers that use longitudinal methodologies study its influence in the chronic phase or once the intensive neurorehabilitation process is completed. There is, therefore, a field to explore in relation to the psychological characteristics of adult patients with moderate-severe acquired brain damage. Furthermore, longitudinal methodology has not been previously used to analyze possible changes in psychological variables during the neurorehabilitation process, nor the influence it may have on its prognosis.

Research Hypothesis:

Psychological characteristics, such as emotional well-being, self-esteem, and motivation, influence neurorehabilitation outcomes in patients with moderate-severe acquired brain damage.

It is expected that:

1. Psychological characteristics associated with greater emotional well-being and psychological adjustment will positively correlate with each other.
2. Demographic, cognitive, and functional indicators will significantly mediate the relationship between psychological characteristics and rehabilitation outcomes.
3. Differences will be observed in psychological characteristics based on the etiology of brain damage, given their varying nature, chronicity, and the neurological sequelae they cause.
4. Trait-type psychological characteristics will remain relatively stable, while state-type characteristics will show significant changes during the neurorehabilitation program.
5. Initial psychological characteristics linked to greater emotional well-being and adjustment will be predictive of better emotional and functional outcomes at the conclusion of the intensive neurorehabilitation process.

Objectives:

To verify the research hypothesis, the following objectives are set:

Main Objective To study the psychological characteristics of individuals with acquired brain damage.

Secondary Objectives:

* SO1: Analyze the relationships among the psychological characteristics studied.
* SO2: Explore the associations between psychological characteristics and other indicators (demographic, cognitive, functional).
* SO3: Investigate differences in psychological characteristics based on the etiology of brain damage.
* SO4: Assess the evolution and changes in psychological characteristics throughout the neurorehabilitation program.
* SO5: Evaluate the prognostic value of initial psychological characteristics in predicting neurorehabilitation outcomes.

Methodology: Prospective observational longitudinal study.

Sample:

After analyzing recent studies that address the same topic, it has been estimated that a sample of approximately 200 participants will be sufficient to meet the proposed objectives.

Inclusion and exclusion criteria are described in the proper section.

Method

Procedure:

At the beginning of the neurorehabilitation program, computerized questionnaires will be administered that assess 14 psychological characteristics (time T1). The same questionnaires will be administered again 2 months later (time T2). In those hospitalized patients who subsequently continue outpatient treatment, a third administration will be carried out 2 months later (time T3).

The 14 selected psychological characteristics will be assessed from 14 standardized questionnaires. The estimated time to complete all the questionnaires is approximately 45 minutes. They will be administered using REDCap (www.project-redcap.org). REDCap is a web application that allows the creation and administration of questionnaires and databases online. Participants will be offered the possibility of completing the questionnaires in person or online. In the second case, the link will be sent to them by email.

The list and characteristics of the main outcome variables are described in its proper section.

Other types of data will also be collected:

* Injury data: NIHHS in the case of patients with stroke, Glasgow Coma Scale in the case of patients with traumatic brain injury.
* Demographic and social data: Age, time since injury, educational level, occupation level, socio-family assessment scale (EVSF-IG).
* Functional data: Functional independence measure (FIM), Barthel index and the gait assessment scale (FAC).
* Measure of therapeutic adherence: Number of the cognitive rehabilitation sessions carried out.
* Cognitive measures:

Orientation: Subtest of orientation in person, space and time of the Barcelona Test (T. B).

Language: Subtest of word repetition, visual-verbal naming and comprehension of orders (T. B).

Gnosis (Visoperception): Subtest of superimposed images (T. B).

Attention:

Attentional span: Digit span (WAIS-III). Selective: TMT-A Divided: TMT-B Sustained: Continuous Performance Test (CPT-3). Verbal memory: Short-term, Long-term, and Recognition (RAVLT).

Executive Functions:

Working memory: Reverse digit span, Letter-Number Sequencing (WAIS-III) Flexibility: PMR, WCST (Perseverative errors). Categorization: WCST (Categories) Visual construction: Block Design (WAIS-III). Processing speed: Digit Symbol(WAIS-III)

Processing of personal data:

All participants will be informed at the beginning of the study of its characteristics, its objectives and the implications of their participation, in order to obtain their consent to participate. For this reason, they will be provided with an information document describing the type of study, the potential advantages and disadvantages, the duration of the project and the procedures that will be applied. In addition, the document will explain very precisely all the measures related to data protection, and the right of participants to decline their participation in the study without consequences, explicitly guaranteeing that there will be no difference in the way in which they may be treated in the future at the center, regardless of their decision to participate in the study; as well as the right to abandon it at any time they consider appropriate, without needing to offer any explanation justifying their decision.

In order to preserve the confidentiality of the subjects who are part of the study, techniques will be used to dissociate personal data from the data that is part of the research object. The researchers will use anonymized data at all times, which they will receive through a query to the IT department from the research and innovation office, who will supervise the effective elimination of any personal data. The procedure will comply at all times with the regulations established in Organic Law 03/2018 of 5 December and Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on Data Protection (GDPR).

Ethical considerations:

* The treatment proposed in the study does not pose any risk to the patients who are part of the sample, while it could be beneficial both for the treatment and for the evaluation of symptoms and functional limitations resulting from brain damage.
* During the study, the international ethical standards for research on humans established in the principles defined in the Declaration of Helsinki and subsequent revisions (Fortalesa, Brazil, October 2013), the code of good clinical practice and national recommendations will be followed in accordance with current legislation established in Law 14/2007 on Biomedical Research.
* Prior to the start of the study, authorization will be requested from the CEIm of the Catalan Union of Hospitals Foundation. Any modification of the protocol, other than administrative changes, will require an amendment to the protocol that will have to be approved by the same Committee.
* The researcher will have to ensure that the participant understands clearly and precisely that his/her participation is voluntary, that it will not affect in any way the way he/she is or may be treated at the center, now or in the future, and that he/she may stop participating at any time, without having to give explanations or justify it.
* The researcher will also explain to each patient the nature of the study, its purposes, procedures, estimated duration, potential risks and benefits related to participation in the study, as well as any inconvenience that this may entail. Each participant will be informed that their participation is voluntary and that they may withdraw from the study at any time, without this affecting their subsequent medical treatment or their relationship with the doctor treating them.
* The patient will have sufficient time to read and understand the researcher's explanations contained in the information sheet (see appendix I) before signing the informed consent (see appendix II). The patient will receive a copy of this document. No patient may be included in the study without first giving written consent.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Present acquired brain damage (stroke, head trauma, encephalopathy, brain tumor, or anoxia) after less than 6 months of evolution.
3. Participants must present a cognitive alteration objectified through a neuropsychological examination.
4. Be correctly oriented in person, space and time (assessed by psychometric tests).
5. Have a good command of Spanish.

   Exclusion Criteria:
6. Presenting a neurological or psychiatric history.
7. Presenting a language disorder or severe visual-perceptive disorder - hemineglect - that prevents participation in the study (does not allow for correct administration of the questionnaire).
8. A posteriori criterion (once the study has begun): Answering incorrectly to any of the validity items included in the questionnaire. This situation leads to automatic exclusion from studies.

The initial neuropsychological examination will be used to check whether participants meet inclusion criteria 3 and 4, as well as exclusion criterion 7. This examination includes orientation tests (subtest of the Barcelona Orientation Test), language tests (subtests of the Barcelona Word Repetition Test, Word Naming and Command Comprehension Test) and visual-perception tests (subtests of the Barcelona Superimposed Figures Test). Only those participants who correctly answer all the items will be selected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who begins neurorehabilitation treatment at the Institut Guttmann Neurorehabilitation Hospital (Badalona) during the recruitment period will be considered a candidate for the study. The inclusion and exclusion criteria will then be checked, and those who meet the criteria will be offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Illness perception | 4 months
  The Brief Illness Perception Questionnaire (BIPQ) 9 items. 1-10 score range for each item. Higher scores describe a higher degree of accord with the correspondent parameter of perception.
Motivation towards rehabilitation | 4 months
  Motivation in stroke patients for rehabilitation scale (MORE)
  17 items. 17-119 score range. Higher scores describe a higher degree of motivation towards rehabilitation.
Personal values | 4 months
  Valued Living Questionnaire - Adapted (22 items) Part A: 11 items. 1-10 score range for each item. Higher scores describe a higher degree of identification towards the specific value.
  Part B: 11 items. 1-4 score range for each item. Higher scores describe a worse perceived impact in the specific value described after the brain injury.
Coping strategies | 4 months
  Coping Orientation to Problems Experienced Inventory - Abbreviated (Brief COPE) 28 items. 28-112 score range. Higher scores describe a higher use of coping strategies.
Depressive symptomatology | 4 months
  Depressive symptomatology measured by Patient Health Questionnaire-9 (PHQ-9) 9 items. 0-27 score range. Higher scores describe higher depressive symptomatology
Anxiety symptomatology | 4 months
  Anxiety symptomatology measured by General Anxiety Disorder Questionnaire (GAD-7) 7 items. 0-21 score range. Higher scores describe higher anxiety symptomatology
Anosognosia | 4 months
  Ad-hoc Anosognosia Questionnaire. 5 Items. 1-20 score range. Higher scores describe a higher perceived cognitive impairment.
Self-Esteem | 4 months
  Rosenberg Self-Esteem scale (RSE) 10 items. 0-30 score range. Higher scores describe a higher degree of Self-Esteem.
Locus of control | 4 months
  Sense of Control Scale. 8 items. 4 subscales with a range of -4 to +4.
  Locus of control refers to the perception of where control lies within their life and the causes of the events.
  A higher "internal good" subscale describes a higher tendency to attribute success towards oneself.
  A higher "external good" subscale describes a higher tendency to attribute success towards elements independent of oneself.
  A higher "internal bad" subscale describes a higher tendency to attribute failure towards oneself.
  A higher "external bad" subscale describes a higher tendency to attribute failure towards elements independent of oneself.
Self-Compassion | 4 months
  Self-Compassion Scale Short Form (SCS-SF) 12 items. 12-60 score range. Higher scores describe a higher degree of Self-Compassion.
Injustice Experience | 4 months
  Injustice Experience Questionnaire; IEQ 12 items. 0-48 score range. Higher scores describe a higher perception of injustice.
Dispositional hope | 4 months
  Life Orientation Test (LOT-R):
  6 items. 0-24 score range. Higher scores describe a higher degree of dispositional hope.
Posttraumatic Growth | 4 months
  Posttraumatic Growth Inventory Short Form (PTGI-SF) 8 items. 0-40 score range. Higher scores describe a higher degree of Posttraumatic Growth.
Personality traits | 4 months
  Big Five Inventory -2 (BFI-2-S) 30 items. 15 subscales with a 2-10 score range. 5 Personality traits with varying ranges of scores. Higher scores describe a higher intensity in that specific personality trait.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Guttmann, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Sharing individual participant data will be considered upon approval by the hospital executive board and ethical committee.

REFERENCES:
- [Background] Chung ML, Bakas T, Plue LD, Williams LS. Effects of Self-esteem, Optimism, and Perceived Control on Depressive Symptoms in Stroke Survivor-Spouse Dyads. J Cardiovasc Nurs. 2016 Mar-Apr;31(2):E8-E16. doi: 10.1097/JCN.0000000000000232. PMID 25658182
- [Background] Yoshida T, Otaka Y, Kitamura S, Ushizawa K, Kumagai M, Yaeda J, Osu R. Influence of motivation on rehabilitation outcomes after subacute stroke in convalescent rehabilitation wards. Front Neurol. 2023 Jul 14;14:1185813. doi: 10.3389/fneur.2023.1185813. eCollection 2023. PMID 37521301
- [Background] Yoshida T, Otaka Y, Kitamura S, Ushizawa K, Kumagai M, Kurihara Y, Yaeda J, Osu R. Development and validation of new evaluation scale for measuring stroke patients' motivation for rehabilitation in rehabilitation wards. PLoS One. 2022 Mar 17;17(3):e0265214. doi: 10.1371/journal.pone.0265214. eCollection 2022. PMID 35298513
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649
- [Background] Sullivan MJ, Adams H, Horan S, Maher D, Boland D, Gross R. The role of perceived injustice in the experience of chronic pain and disability: scale development and validation. J Occup Rehabil. 2008 Sep;18(3):249-61. doi: 10.1007/s10926-008-9140-5. Epub 2008 Jun 7. PMID 18536983
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Soto CJ, John OP. The next Big Five Inventory (BFI-2): Developing and assessing a hierarchical model with 15 facets to enhance bandwidth, fidelity, and predictive power. J Pers Soc Psychol. 2017 Jul;113(1):117-143. doi: 10.1037/pspp0000096. Epub 2016 Apr 7. PMID 27055049
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Martin-Albo J, Nuniez JL, Navarro JG, Grijalvo F. The Rosenberg Self-Esteem Scale: translation and validation in university students. Span J Psychol. 2007 Nov;10(2):458-67. doi: 10.1017/s1138741600006727. PMID 17992972
- [Background] Rodero B, Luciano JV, Montero-Marin J, Casanueva B, Palacin JC, Gili M, Lopez del Hoyo Y, Serrano-Blanco A, Garcia-Campayo J. Perceived injustice in fibromyalgia: psychometric characteristics of the Injustice Experience Questionnaire and relationship with pain catastrophising and pain acceptance. J Psychosom Res. 2012 Aug;73(2):86-91. doi: 10.1016/j.jpsychores.2012.05.011. Epub 2012 Jun 20. PMID 22789409
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Pacheco-Huergo V, Viladrich C, Pujol-Ribera E, Cabezas-Pena C, Nunez M, Roura-Olmeda P, Amado-Guirado E, Nunez E, Del Val JL; en representacion del Grupo IPQ-R. [Perception in chronic illnesses: linguistic validation of the revised Illness Perception Questionnaire and the Brief Illness Perception Questionnaire for a Spanish population]. Aten Primaria. 2012 May;44(5):280-7. doi: 10.1016/j.aprim.2010.11.022. Epub 2011 Sep 28. Spanish. PMID 21955598
- [Background] Nakamori M, Imamura E, Tachiyama K, Kamimura T, Hayashi Y, Matsushima H, Okamoto H, Mizoue T, Wakabayashi S. Patient Health Questionnaire-9 predicts the functional outcome of stroke patients in convalescent rehabilitation ward. Brain Behav. 2020 Dec;10(12):e01856. doi: 10.1002/brb3.1856. Epub 2020 Sep 20. PMID 32951302
- [Background] Miller LR, Divers R, Reed C, Cherry J, Patrick A, Calamia M. Value-consistent rehabilitation is associated with long-term psychological flexibility and quality of life after traumatic brain injury. Neuropsychol Rehabil. 2024 Aug;34(7):955-973. doi: 10.1080/09602011.2023.2256964. Epub 2023 Sep 14. PMID 37708399
- [Background] McIntyre A, Mehta S, Janzen S, Rice D, Harnett A, MacKenzie HM, Vanderlaan D, Teasell R. Coping strategies and personality traits among individuals with brain injury and depressive symptoms. NeuroRehabilitation. 2020;47(1):25-34. doi: 10.3233/NRE-203081. PMID 32675425
- [Background] Martinez-Vazquez S, Martinez-Galiano JM, Peinado-Molina RA, Gutierrez-Sanchez B, Hernandez-Martinez A. Validation of General Anxiety Disorder (GAD-7) questionnaire in Spanish nursing students. PeerJ. 2022 Nov 1;10:e14296. doi: 10.7717/peerj.14296. eCollection 2022. PMID 36340193
- [Background] Leventhal H, Phillips LA, Burns E. The Common-Sense Model of Self-Regulation (CSM): a dynamic framework for understanding illness self-management. J Behav Med. 2016 Dec;39(6):935-946. doi: 10.1007/s10865-016-9782-2. Epub 2016 Aug 11. PMID 27515801
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Groeneveld IF, van der Pas SL, Meesters JJL, Schuurman JM, van Meijeren-Pont W, Jagersma E, Goossens PH, Kaptein AA, Vliet Vlieland TPM; SCORE-study group. Illness perceptions of stroke survivors: Predictors and changes over time - A 1 year follow-up study. J Psychosom Res. 2019 Jan;116:54-61. doi: 10.1016/j.jpsychores.2018.10.019. Epub 2018 Nov 2. PMID 30654994
- [Background] Garrido-Hernansaiz H, Rodriguez-Rey R, Collazo-Castineira P, Collado S. The posttraumatic growth inventory-short form (PTGI-SF): A psychometric study of the spanish population during the COVID-19 pandemic. Curr Psychol. 2022 Jan 11:1-10. doi: 10.1007/s12144-021-02645-z. Online ahead of print. PMID 35035195
- [Background] Garcia-Campayo J, Navarro-Gil M, Andres E, Montero-Marin J, Lopez-Artal L, Demarzo MM. Validation of the Spanish versions of the long (26 items) and short (12 items) forms of the Self-Compassion Scale (SCS). Health Qual Life Outcomes. 2014 Jan 10;12:4. doi: 10.1186/1477-7525-12-4. PMID 24410742
- [Background] Diez-Quevedo C, Rangil T, Sanchez-Planell L, Kroenke K, Spitzer RL. Validation and utility of the patient health questionnaire in diagnosing mental disorders in 1003 general hospital Spanish inpatients. Psychosom Med. 2001 Jul-Aug;63(4):679-86. doi: 10.1097/00006842-200107000-00021. PMID 11485122
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744